CLINICAL TRIAL: NCT02234622
Title: Outcomes of a Holistic Yoga Program Designed to Relieve PTSD (RELIEVE Trial)
Brief Title: Comparing Effects of a Holistic Yoga Program and a Wellness Program on PTSD Symptoms
Acronym: RELIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1487-R
Record Dates: First submitted 2014-08-29; First posted 2014-09-09 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Stress Disorders, Post-Traumatic; Yoga; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Holistic Yoga Program (Experimental): The Holistic Yoga Program (HYP) (postures, breathing practices, deep muscle contraction practices, relaxation) is a 16 week, 90 minute weekly group intervention.
  Interventions: Behavioral: Holistic Yoga Program
- Wellness Lifestyle Program (Active Comparator): The Wellness Lifestyle Program (WLP) is a 16 week, 90 minute weekly group intervention consisting of low intensity walking with didactics about wellness topics.
  Interventions: Behavioral: Wellness Lifestyle Program

INTERVENTIONS:
Behavioral: Holistic Yoga Program — The Holistic Yoga Program (HYP) (postures, breathing practices, deep muscle contraction practices, relaxation) is a 16 week, 90 minute weekly group intervention.
  Other Names: HYP
  Arms: Holistic Yoga Program
Behavioral: Wellness Lifestyle Program — The Wellness Lifestyle Program (WLP) is a 16 week, 90 minute weekly group intervention consisting of low intensity walking with didactics about wellness topics.
  Other Names: WLP
  Arms: Wellness Lifestyle Program

SUMMARY:
Given the limited effectiveness of current treatments and the burden PTSD places on Veterans, civilians and clinicians, this research aims to compare the effects of a standardized, traditional, holistic yoga intervention (postures, breathing, deep muscle contraction and relaxation practices) with a wellness program (wellness topics and physical activity) on PTSD symptoms.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder constitutes a substantial proportion of the burden of illness among Veterans. However, current PTSD treatments are not effective for all, and a significant number remain symptomatic despite pharmacotherapy and psychotherapy. As a result, there has been increased interest within the military and VA in Complementary and Alternative Medicine approaches, such as yoga, to improve symptoms without requiring direct verbal processing of the trauma. Yoga provides an innovative approach to calming hyperarousal, reducing numbness/avoidance, and improving self-regulation of emotions, while cultivating physical and emotional well-being. Because of this unique approach to the biological, psychological, and social dimensions of PTSD, we believe that yoga interventions are poised to meet the demand for more effective PTSD treatment options for Veterans. Recent research indicates that yoga interventions can be delivered successfully to individuals who have PTSD and have the potential to reduce clinician rated and self-reported overall PTSD symptoms, depression and anxiety. However, few studies exist that have evaluated yoga for PTSD and they have involved small sample sizes and are either uncontrolled or waitlist/usual care controlled. Also, there is much variation among studies in the style and components of yoga interventions. Thus, a randomized controlled trial of a standardized, traditional, holistic yoga intervention is urgently needed to inform VA policy makers and clinicians of the potential benefits of yoga as an adjunct to currently available PTSD treatments.

OBJECTIVE: The overall goal of this project is to compare the effects of a 16-week Holistic Yoga Program (HYP) with a 16-week Wellness Lifestyle Program (WLP) on PTSD and related symptoms and outcomes. This project has three specific aims: 1) to compare the effects of the interventions (HYP vs. WLP) on overall PTSD symptom severity; 2) compare the interventions' effects on PTSD-specific symptoms (anger, sleep), PTSD-related symptoms (depression, anxiety, pain) and related outcomes (well-being/quality of life); 3) to manualize the Holistic Yoga Program and training process for experienced yoga teachers to deliver HYP to individuals who have PTSD in order to facilitate future study and dissemination efforts.

METHODS: This study sample will include 212 outpatients with a clinician-confirmed diagnosis of PTSD, recruited from the Roudebush VA Medical Center as well as metropolitan area mental health clinicians and military/Veterans' organizations, who will be randomly assigned to receive the Holistic Yoga Program (HYP) or the Wellness Lifestyle Program (WLP). The HYP will involve a standardized 16-week intervention consisting of: 1) in-person group yoga class taught by a yoga therapist (Yoga Alliance minimum 200 hour level) with trained assistants.Classes will include (1) yoga postures, breathing practices, deep muscle contraction practices, relaxation practices, and integration of scientific rational and yoga philosophy within the instruction; (2) video and audio recordings for home practice; and 4) a Participant Handbook to reinforce concepts taught during in-person sessions. The WLP is an attention control comprised of low intensity walking and didactics about wellness topics that will also encourage home practice and provide a Participant Handbook to reinforce concepts taught during in-person sessions.

ELIGIBILITY:
Inclusion Criteria:

Veterans and civilians will be eligible for inclusion if

* they are age 18 or older,
* have a Clinician Administered PTSD Scale-confirmed PTSD diagnosis,
* and access to a working telephone for ease of contact during the course of the study.

Exclusion Criteria:

Exclusion criteria will include:

* severe medical conditions in which yoga is contraindicated;
* active psychosis;
* active suicidal intent;
* moderate to severe cognitive impairment as determined by the short Mini-Mental State Examination, a six-item screener (MMSE);
* involvement in ongoing yoga classes and/or regular home practice of yoga in the previous 3 months;
* and receiving ongoing medical or psychological treatment that includes more than one hour weekly of relaxation and mind-body based stress reduction strategies (related directly to meditation and yoga).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louanne W Davis, PsyD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wellness Lifestyle Program: The Wellness Lifestyle Program (WLP) is a 16 week, 90 minute weekly group intervention consisting of low intensity physical activity with didactics about wellness topics.
  Wellness Lifestyle Program: The Wellness Lifestyle Program (WLP) is a 16 week, 90 minute weekly group intervention consisting of low intensity physical activity (walking) with didactics about wellness topics.
Period: Overall Study
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
Started | 108 | 104
Completed | 65 | 68
Not Completed | 43 | 36
Not completed — Withdrawal by Subject | 16 | 22
Not completed — Lost to Follow-up | 27 | 14

BASELINE CHARACTERISTICS:
Population: three participants were removed from the analysis when results of a retrospective audit of baseline PTSD diagnosis indicated they did not meet diagnostic criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program | Total
Number analyzed (Participants) | 108 | 101 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (12.6) | 51.2 (13.3) | 50.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 71
  Male | 70 | 68 | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 32 | 33 | 65
  White | 69 | 60 | 129
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 108 | 101 | 209
Clinician Administered PTSD Scale 5 [Mean (Standard Deviation); unit: units on a scale] — Scores range 0-80 with higher scores meaning a worse outcome.
  units on a scale | 37.1 (8.7) | 36.0 (8.7) | 36.57 (8.71)
PTSD Checklist 5 [Mean (Standard Deviation); unit: units on a scale] — Scores range 0-80 with higher scores indicating worse outcome.
  units on a scale | 45.2 (12.1) | 45.1 (13.0) | 45.14 (12.51)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS-5)
Description: The CAPS is a semi-structured clinician administered interview that measures PTSD diagnostic status and symptom severity consistent with the Diagnostic and Statistical Manual-Fifth Edition. Scores range 0-80 with higher scores meaning a worse outcome.
Time Frame: Change from baseline to 16 weeks (end of treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Wellness Lifestyle Program: The Wellness Lifestyle Program (WLP) is a 16 week, 90 minute weekly group intervention consisting of low intensity physical activity with didactics about wellness topics.
  Wellness Lifestyle Program: The Wellness Lifestyle Program (WLP) is a 16 week, 90 minute weekly group intervention consisting of low intensity physical activity with didactics about wellness topics.
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
Number analyzed (Participants) | 108 | 101
score on a scale | 25.8 (12.1) | 31.0 (13.0)
Statistical Analysis 1: Comparison: Holistic Yoga Program vs Wellness Lifestyle Program; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-8.2 to -1.8], Standard Error of Mean 1.6

2. Primary Outcome: PTSD Checklist
Description: PTSD self-reported symptom severity will be assessed with the PTSD Checklist-5 (PCL-5), a 20-item self-report measure of the 5th version of the Diagnostic and Statistics Manual (DSM-5) symptoms of PTSD used as a measure of change in PTSD symptoms as a function of treatment. Scores range 0-80 with higher scores indicating worse outcome.
Time Frame: Change from baseline to 16 weeks (end of treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
Number analyzed (Participants) | 108 | 101
score on a scale | 33 (17.5) | 40.2 (15.2)
Statistical Analysis 1: Comparison: Holistic Yoga Program vs Wellness Lifestyle Program; Test type: Superiority; p = 0.005, Mixed Models Analysis; Mean Difference (Net) = -6.1, 95% CI 2-sided [-10.3 to -1.8], Standard Error of Mean 2.2

3. Secondary Outcome: Medical Outcomes Study 12-item Sleep Scale (MOS) Problem Index II
Description: Medical Outcomes Study Sleep Scale (MOS) Problem Index II is a 9-item sub-scale of the 12-item MOS self-report measure that assesses sleep quality (sleep disturbance, adequacy of sleep, and sleep quantity). The item scores of the 9-item sub-scale range from 1-6 and the sub-scale totals are converted to scores ranging 0-100, with higher scores indicating a worse outcome.
Time Frame: Change from baseline to 16 weeks (end of treatment)
Population: three participants were removed from the analysis when a retrospective audit of the Clinician Administered PTSD Scale revealed they did not meet diagnostic criteria for PTSD
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
Number analyzed (Participants) | 108 | 101
score on a scale | 45 (21.2) | 55 (20.7)
Statistical Analysis 1: Comparison: Holistic Yoga Program vs Wellness Lifestyle Program; Test type: Superiority; p = 0.042, Mixed Models Analysis; Mean Difference (Final Values) = -6.7, 95% CI 2-sided [-11.9 to -1.6], Standard Error of Mean 2.6

4. Secondary Outcome: Patient Reported Outcome Measure Information System (PROMIS) - Short Form 5a
Description: PROMIS - short form 5a is a 5-item self-report measure to assess feelings of anger over the past 7 days. Total scores, ranging 5-25 are converted to T-scores with higher scores indicating poorer outcome. A score of 50 represents the mean. A difference of 10 from the mean indicates a difference of one standard deviation. Thus, a score of 60 is one standard deviation above the mean, while a score of 30 is two standard deviations below the mean. T-scores range from 0-100
Time Frame: Change from baseline to 16 weeks (end of treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
Number analyzed (Participants) | 108 | 101
score on a scale | 57.1 (8.9) | 58.9 (9.2)
Statistical Analysis 1: Comparison: Holistic Yoga Program vs Wellness Lifestyle Program; Test type: Superiority; p = 0.482, Mixed Models Analysis; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.2 to 1.1], Standard Error of Mean 1.4

5. Secondary Outcome: Beck Depression Inventory-II
Description: Depression will be measured by the Beck Depression Inventory (BDI), a 21-item self-report measure, the total score of which ranges 0-63 with higher scores indicating a poorer outcome.
Time Frame: Change from baseline to 16 weeks (end of treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
Number analyzed (Participants) | 108 | 101
score on a scale | 17.4 (12.2) | 18.7 (10.7)
Statistical Analysis 1: Comparison: Holistic Yoga Program vs Wellness Lifestyle Program; Test type: Superiority; p = 0.635, Mixed Models Analysis; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-4.7 to 1.9], Standard Error of Mean 1.7

6. Secondary Outcome: Spielberger State-Trait Anxiety (STAI) - State Subscale
Description: Anxiety will be measured by the Spielberger State-Trait Anxiety Inventory (STAI), State Anxiety subscale, a self-report instrument consisting of 20-items rated on a 4-point scale (1-4), with a possible range of 20-80. Higher scores indicate worse outcome.
Time Frame: Change from baseline to 16 weeks (end of treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
Number analyzed (Participants) | 108 | 101
score on a scale | 29.5 (11) | 27.6 (11.6)
Statistical Analysis 1: Comparison: Holistic Yoga Program vs Wellness Lifestyle Program; Test type: Superiority; p = 0.367, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-6.0 to 1.1], Standard Error of Mean 1.8

7. Secondary Outcome: Brief Pain Inventory (BPI) Item #3
Description: Pain will be assessed using the Brief Pain Inventory (BPI), item #3 which is an indicator of average pain severity in the past week. Scores range from 0-10 with higher scores indicating poorer outcome.
Time Frame: Change from baseline to 16 weeks (end of treatment)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
Number analyzed (Participants) | 108 | 101
score on a scale | 4.9 (2.7) | 4.9 (2.9)
Statistical Analysis 1: Comparison: Holistic Yoga Program vs Wellness Lifestyle Program; Test type: Superiority; p = 0.668, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.0], Standard Error of Mean 0.4

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Holistic Yoga Program | Wellness Lifestyle Program
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/104
Other Adverse Events (participants affected / at risk) | 0/108 | 0/104

LIMITATIONS AND CAVEATS:
All participants were from one large city in the Midwest. The yoga intervention was designed to address PTSD by a yoga therapist who trained the yoga teacher assistants and may not apply to all types of yoga classes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT02234622/Prot_SAP_000.pdf